CLINICAL TRIAL: NCT05901857
Title: Assessing the Precision of Convolutional Neural Networks for Dental Age Estimation in an Egyptian Population From Digital Panoramic Radiographs: A Diagnostic Accuracy Study
Brief Title: Assessing the Precision of Convolutional Neural Networks for Dental Age Estimation From Panoramic Radiographs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rawan Abdel Wahhab Bahaa Eldin Elkassas, Principal Investigator, Cairo University
Other Study IDs: ORAD 3-3-1 (2)
Record Dates: First submitted 2023-05-12; First posted 2023-06-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Age Problem
MeSH Terms: interventions — Convolutional Neural Networks

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: convolutional neural network — A deep learning model for dental age classification from panoramic images

SUMMARY:
The aim of this study is to assess the accuracy of a convolutional neural network in dental age estimation from digital panoramic radiographs. The reference standard will be the chronological age of the patient.

DETAILED DESCRIPTION:
Willems method is a dental age estimation technique modiﬁed from Demirjian method by creating new tables from which a maturity score is directly expressed in years.

Panoramic radiographs of all participants will be taken with their informed consent, then they will be numbered and coded. Chronological age for each participant will be calculated by subtracting date of birth from date of radiograph and the real age will be blinded from the researcher (The chronological age is the ground truth). All panoramic radiographs will be examined twice by the main author to determine the dental age according to Willems method.

The seven mandibular left teeth excluding the third molar will be scored as '0' for absence of calcification, and 'A' to 'H', depending on the stage of calcification. Each letter corresponds to a score which is the dental age fraction using tables for boys and girls. Summing the scores for the seven left mandibular teeth directly will result in the estimated dental age. The dental radiologist estimation accurancy will be compared to the ground truth (first index test).

The second index test which will also be compared to the ground truth is the CNN model. To prepare the dataset for the CNN model, a rigorous preprocessing procedure will be followed. This will involve resizing the images to the desired dimensions, segmenting the teeth parts to be included in the image, and applying data augmentation techniques to enhance the quality and quantity of the dataset. The dataset will then be split into training and testing sets using a 20:80 ratio, which will be carefully selected based on the expected number of samples. Also the accuracy of the model will be assessed compared to the ground truth (the chronological ages).

ELIGIBILITY:
Inclusion Criteria:

* Presence of all mandibular left permanent teeth (except third molars)
* Clearly visible root development
* No systemic disease
* No history of root canal therapy or extraction
* No related diseases affecting mandibular development such as cysts or tumors.

Exclusion Criteria:

* Patients with premature birth
* Facial asymmetry
* Congenital anomalies
* History of trauma or surgery in dentofacial region

Ages: 6 Years to 16 Years | Sex: All
Age Groups: Child
Study Population: Panoramic radiographs will be recruited from Faculty of Dentistry, Oral Radiology Department.
Sampling Method: Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2023-06-30 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of dental age estimation from digital panoramic radiographs using CNN models | Through study completion, an average of 1 year
  Percentage

CONTACTS AND LOCATIONS:
Overall Officials: Mohab Eid, Study Chair — Nile University
Locations (1):
- Rawan Elkassas, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Banar N, Bertels J, Laurent F, Boedi RM, De Tobel J, Thevissen P, Vandermeulen D. Towards fully automated third molar development staging in panoramic radiographs. Int J Legal Med. 2020 Sep;134(5):1831-1841. doi: 10.1007/s00414-020-02283-3. Epub 2020 Apr 1. PMID 32239317
- [Background] Ekert T, Krois J, Meinhold L, Elhennawy K, Emara R, Golla T, Schwendicke F. Deep Learning for the Radiographic Detection of Apical Lesions. J Endod. 2019 Jul;45(7):917-922.e5. doi: 10.1016/j.joen.2019.03.016. Epub 2019 Jun 1. PMID 31160078
- [Background] El-Desouky SS, Kabbash IA. Age estimation of children based on open apex measurement in the developing permanent dentition: an Egyptian formula. Clin Oral Investig. 2023 Apr;27(4):1529-1539. doi: 10.1007/s00784-022-04773-7. Epub 2022 Nov 17. PMID 36394611
- [Background] Galibourg A, Cussat-Blanc S, Dumoncel J, Telmon N, Monsarrat P, Maret D. Comparison of different machine learning approaches to predict dental age using Demirjian's staging approach. Int J Legal Med. 2021 Mar;135(2):665-675. doi: 10.1007/s00414-020-02489-5. Epub 2021 Jan 7. PMID 33410925
- [Background] Guo YC, Han M, Chi Y, Long H, Zhang D, Yang J, Yang Y, Chen T, Du S. Accurate age classification using manual method and deep convolutional neural network based on orthopantomogram images. Int J Legal Med. 2021 Jul;135(4):1589-1597. doi: 10.1007/s00414-021-02542-x. Epub 2021 Mar 4. PMID 33661340
- [Background] Kim S, Lee YH, Noh YK, Park FC, Auh QS. Age-group determination of living individuals using first molar images based on artificial intelligence. Sci Rep. 2021 Jan 13;11(1):1073. doi: 10.1038/s41598-020-80182-8. PMID 33441753
- [Background] Sehrawat JS, Singh M. Willems method of dental age estimation in children: A systematic review and meta-analysis. J Forensic Leg Med. 2017 Nov;52:122-129. doi: 10.1016/j.jflm.2017.08.017. Epub 2017 Aug 25. PMID 28918371
- [Background] Shen S, Liu Z, Wang J, Fan L, Ji F, Tao J. Machine learning assisted Cameriere method for dental age estimation. BMC Oral Health. 2021 Dec 15;21(1):641. doi: 10.1186/s12903-021-01996-0. PMID 34911516
- [Background] Vila-Blanco N, Carreira MJ, Varas-Quintana P, Balsa-Castro C, Tomas I. Deep Neural Networks for Chronological Age Estimation From OPG Images. IEEE Trans Med Imaging. 2020 Jul;39(7):2374-2384. doi: 10.1109/TMI.2020.2968765. Epub 2020 Jan 31. PMID 32012002
- [Background] Ye X, Jiang F, Sheng X, Huang H, Shen X. Dental age assessment in 7-14-year-old Chinese children: comparison of Demirjian and Willems methods. Forensic Sci Int. 2014 Nov;244:36-41. doi: 10.1016/j.forsciint.2014.07.027. Epub 2014 Aug 19. PMID 25195126